CLINICAL TRIAL: NCT03460886
Title: Most Effective Stimulation Site in Transcranial Direct Current Stimulation for Gait Recovery After Stoke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-11-080
Record Dates: First submitted 2018-01-22; First posted 2018-03-09 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Stroke; Gait Disorders, Neurologic
Keywords: transcranial direct current stimulation
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bihemispheric stimulation (Experimental): 1. Anodal stimulation on ipsilesional leg motor primary cortex and supplementary motor area
  2. Anodal stimulation on contralesional leg motor primary cortex and supplementary motor area Subject walks on treadmill for 10 minute during stimulation.
  Interventions: Device: Ipsilesional stimulation; Device: Contralesional stimulation; Other: Walking on treadmill
- Ipsilesional stimulation (Experimental): 1. Anodal stimulation on ipsilesional leg motor primary cortex and supplementary motor area
  2. Sham on contralesional leg motor primary cortex and supplementary motor area Subject walks on treadmill for 10 minute during stimulation.
  Interventions: Device: Ipsilesional stimulation; Other: Walking on treadmill
- Contralesional stimulation (Experimental): 1. Sham stimulation on ipsilesional leg motor primary cortex and supplementary motor area
  2. Anodal stimulation on contralesional leg motor primary cortex and supplementary motor area Subject walks on treadmill for 10 minute during stimulation.
  Interventions: Device: Contralesional stimulation; Other: Walking on treadmill
- Sham (Active Comparator): 1. Sham stimulation on ipsilesional leg motor primary cortex and supplementary motor area
  2. Sham stimulation on contralesional leg motor primary cortex and supplementary motor area Subject walks on treadmill for 10 minute during stimulation.
  Interventions: Other: Walking on treadmill

INTERVENTIONS:
Device: Ipsilesional stimulation — anodal stimulation on Ipsilesional leg area of primary motor cortex and supplementary motor area for 30 minutes
  Arms: Bihemispheric stimulation; Ipsilesional stimulation
Device: Contralesional stimulation — anodal stimulation on contralesional leg area of primary motor cortex and supplementary motor area for 30 minutes
  Arms: Bihemispheric stimulation; Contralesional stimulation
Other: Walking on treadmill — walking on treadmill for 10 minutes

SUMMARY:
The aim of this study is to investigate the most effective stimulation site in transcranial direct current stimulation for gait recovery after stroke. All subjects will go through four conditions of transcranial direct current stimulation with for 30 minutes. Four conditions are 1) bihemispheric stimulation - anodal stimulation on both ipsilesional and contralesional leg area of primary motor cortex and supplementary motor area. 2) ipsilesional stimulation - anodal stimulation on ipsilesional leg area of primary motor cortex and supplementary motor area. 3) contralesional stimulation - anodal stimulation on contralesional leg area of primary motor cortex and supplementary motor area. 4) sham stimulation. Subjects will walk on treadmill for 10 minutes during transcranial direct current stimulation. Motor evoked potential and functional evaluations will be done before and after stimulation to measure the changes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients with 6 months after onset.
* Functional ambulation category ≥ 3

Exclusion Criteria:

* patients who needs assist in surface level walking
* patients with mini mental status exam score under 9
* patients with implantable electronic device
* metal device inside skull
* history of epilepsy
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in motor evoked potential | before and after intervention (approximately 30 minutes)
  measure the motor threshold and amplitude of motor evoked potential in tibialis anterior muscle.

SECONDARY OUTCOMES:
Changes in motricity index | before and after intervention (approximately 30 minutes)
  measures motor function
Changes in Fugl Meyer Assessment | before and after intervention (approximately 30 minutes)
  Fugl Meyer Assessment is a measurement of motor function.
Changes in 10 meter walking test | before and after intervention (approximately 30 minutes)
  measures gait speed
Timed up and go test | before and after intervention (approximately 30 minutes)
  measures gait capacity and balance
Functional ambulatory category | before and after intervention (approximately 30 minutes)
  measure gait ability. 0 is impossible to gait and 6 is normal.
Modified ashworth scale | before and after intervention (approximately 30 minutes)
  measures spasticity with scale from 0 to 3. 0 is no increase in muscle tone. 3 is considerable increase in muscle tone, passive movement difficult.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No